CLINICAL TRIAL: NCT04065776
Title: A Phase II Study of Hippocampal-Avoidance Using Proton Therapy in Low-Grade Glioma
Brief Title: Evaluation of Hippocampal-Avoidance Using Proton Therapy in Low-Grade Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HALGG
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Glioma; Pilocytic Astrocytoma; Pilomyxoid Astrocytoma; Pleomorphic Xanthoastrocytoma; Ganglioglioma; Optic Pathway Glioma; Diffuse Astrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma; Ganglioglioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hippocampal-avoidance proton therapy (Experimental): Hippocampal-avoidance proton therapy
  Interventions: Radiation: Hippocampal-avoidance proton therapy

INTERVENTIONS:
Radiation: Hippocampal-avoidance proton therapy — Hippocampal-avoidance proton therapy

SUMMARY:
Low-grade gliomas (LGGs) are the most common brain tumors in children, and a subset of these tumors are treated definitively with focal radiation therapy (RT). These patients often survive for many years after receiving RT and experience late deficits in memory. Verbal recall is an important measure of memory and is associated with other important functional outcomes, such as problem-solving, independence of every-day functioning, and quality of life. Decline in memory, as measured by verbal recall, is associated with RT dose to the hippocampi. Therefore, this phase II study investigates the feasibility of reducing RT doses to the hippocampi (i.e., hippocampal avoidance [HA]) by using proton therapy for midline or suprasellar LGGs.

Primary Objective:

* To determine the feasibility of HA with proton therapy in suprasellar or midline LGGs. Feasibility will be established if 70% of plans meet the first or second dose constraints shown below.

  1. First priority RT dose constraints for bilateral hippocampi: volume receiving 40 CGE (V40CGE) ≤ 25%, dose to 100% of Hippocampus (D100%) ≤ 5CGE.
  2. Second priority RT dose constraints for bilateral hippocampi: V40CGE ≤ 35%, D100% ≤ 10 CGE.

     Secondary Objectives:
* To estimate the 3-year event-free-survival (EFS) for LGGs treated with HA.
* To estimate the change in California Verbal Learning Test short-term delay (CVLT-SD) from baseline to 3 years and from baseline to 5 years
* To compare CVLT-SD and Cogstate neurocognitive scores in patients with proton therapy plans that: (1) meet first priority RT dose constraints, (2) meet second priority RT dose constraints but not first priority RT dose constraints, and (3) that did not meet either first or second RT priority dose constraints

Exploratory Objectives:

* To describe the change in overall cognitive performance from baseline to 3 years and from baseline to 5 years with an age appropriate battery, including gold standard measures shown in the published studies to be sensitive to attention, memory processing speed and executive function that will afford comparison to historical controls.
* To characterize longitudinal changes in connection strength within brain networks in the first 3 years after proton therapy and to investigate associations between these changes and neurocognitive performance with focus on the hippocampi.
* To correlate the distribution and change in L-methyl-11C-methionine positron emission tomography (MET-PET) uptake to tumor progression and from baseline to 3 years and to investigate whether cases of pseudoprogression exhibit a differential pattern of uptake and distribution compared to cases of true progression after controlling for histology.
* To investigate the effect of BRAF alteration, tumor histology and tumor location on PFS and OS in a prospective cohort of patients treated in a homogenous manner.
* To investigate whether the methylation profiles of LGGs differ by tumor location (thalamic/midbrain vs. hypothalamic/optic pathway vs. others) and histologies (pilocytic astrocytoma vs. diffuse astrocytoma vs. others), which, in conjunction with specific genetic alterations, may stratify patients into different subgroups and highlight different therapeutic targets.
* To record longitudinal measures of circulating tumor DNA (ctDNA) in plasma and correlate these measures with radiographic evidence of disease progression.
* To bank formalin-fixed, paraffin-embedded (FFPE)/frozen tumors and whole blood from subjects for subsequent biology studies not currently defined in this protocol.
* To quantify and characterize tumor infiltrating lymphocytes (TILs) and to characterize the epigenetics of T cells and the T cell receptor repertoire within the tumor microenvironment.
* To estimate the cumulative incidence of endocrine deficiencies, vision loss, hearing loss and vasculopathy after proton therapy and compare these data to those after photon therapy.

DETAILED DESCRIPTION:
All patients will receive HA proton therapy to 52.2 CGE or 54 CGE in 29 or 30 fractions, depending on tumor location. Patients will receive weekly magnetic resonance imaging (MRI) scans during the course of proton therapy to monitor changes in solid tumor or cystic volume. Such changes may prompt adaptive therapy to improve coverage or minimize the RT dose to healthy structures. Neurocognitive outcomes, sensitive to measures of memory and learning, will be collected at baseline and continue to 5 years post therapy. Disease evaluation will be monitored with brain MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of pilocytic astrocytoma, pilomyxoid astrocytoma, pleomorphic xanthoastrocytoma, ganglioglioma, optic pathway glioma, diffuse astrocytoma, low-grade neuroepithelial tumor, low-grade glioneuronal tumor or LGG, or not otherwise specified (NOS).
* Patient with eligible diagnosis other than optic pathway glioma or tumors of the brainstem/midbrain/tectum has histologic verification of disease at diagnosis or recurrence OR
* Patient with optic pathway glioma or tumors of the brainstem/midbrain/tectum has radiologic verification of disease at diagnosis or recurrence
* A repeat biopsy was done because the recurrent tumor was enhancing but did not originally enhance because there was a high index of suspicion regarding high-grade transformation
* Tumor must be located in the suprasellar region or midline structures. Midline structures include, but are not limited to, the thalamus, basal ganglia, internal capsule, midbrain, tectum, third ventricle, fourth ventricle, cerebellum, pons, and medulla. Tumors may involve the optic pathway. For questions about tumor locations that are not specified on this list, please contact the Study PI.
* Patients must be at least 6 years but less than 22 years of age at the time of enrollment.
* Patients must have a performance status greater or equal to 70 (use Karnofsky scale for patients aged 16 years and older and Lansky scale for patients aged less than 16 years).
* Patients may not receive concurrent chemotherapy or targeted therapy, including but not limited to BRAF-inhibitors and MEK-inhibitors.
* All patients must be able to undergo contrast-enhanced brain MRI.
* All patients must have adequate organ function as described below.

  * Peripheral absolute neutrophil count (ANC) ≥ 1000/µL
  * Platelet count ≥ 10,000/µL (transfusion independent)
  * Patients with seizures may be enrolled if well controlled on anticonvulsants

Exclusion Criteria:

* Patients may not have received prior CNS radiation.
* Patients with gross total resection and no measurable disease via MRI are not eligible. Patients must have measurable disease of at least 1 cm via MRI.
* Patients with evidence of metastatic disease are not eligible.
* Patients with WHO grade II midline tumors that harbor the H3K27M mutation, IDH-mutant gliomas, grade II ependymomas and subependymomas, pituicytomas, spindle cell oncocytomas, or granular cell tumors of the sellar region are not eligible.
* Patients with tumors that directly invade the hippocampus or with gross tumor volumes that extend into the hippocampus are not eligible.
* Patients with tumors in the spine or cervicomedullary junction.
* Females of child-bearing potential cannot be pregnant or breast feeding. Female participants > 10 years of age or post menarche must have a negative serum or urine pregnancy test before enrollment. Males and females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Patients who are status post resection of bilateral hippocampi. Patients who are status post resection of one hippocampus will be eligible for the study and the hippocampal dose constraints will be applied to the intact hippocampus.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of plans meet the first or second dose constraints. | 4 years after activation
  To determine the feasibility of HA with proton therapy in suprasellar or midline LGGs. Feasibility will be established if 70% of plans meet the first or second dose constraints. First RT dose constraints for bilateral hippocampi: volume receiving 40 CGE (V40CGE) ≤ 25%, dose to 100% of hippocampus (D100%) ≤ 5CGE. Second RT dose constraints for bilateral hippocampi: V40CGE ≤ 35%, D100% ≤ 10 CGE.

SECONDARY OUTCOMES:
EFS of LGGs treated with HA | 3 years
  EFS will be calculated from the date of RT starts until disease progression, second malignancy, death of any cause or last follow up date.
The change in CVLT-SD scores from baseline to 3 years | Baseline evaluation date, 3 years after treatment
  CVLT-SD scores change of patients with HA feasible from baseline evaluation date to 3 years after treatment
The change in CVLT-SD scores from baseline to 5 years | Baseline evaluation date, 5 years after treatment
  CVLT-SD scores change from baseline evaluation date to 5 years after treatment
Cogstate neurocognitive scores | Baseline evaluation date
  Cogstate neurocognitive scores in patients with proton therapy plans
Cogstate neurocognitive scores | 3 years after treatment
  Cogstate neurocognitive scores in patients with proton therapy plans
Cogstate neurocognitive scores | 5 years after treatment
  Cogstate neurocognitive scores in patients with proton therapy plans
CVLT-SD neurocognitive scores | Baseline evaluation date
  CVLT-SD neurocognitive scores in patients with proton therapy plans
CVLT-SD neurocognitive scores | 3 years after treatment
  CVLT-SD neurocognitive scores in patients with proton therapy plans
CVLT-SD neurocognitive scores | 5 years after treatment
  CVLT-SD neurocognitive scores in patients with proton therapy plans

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Merchant, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols